CLINICAL TRIAL: NCT02474433
Title: Same-day Cervical Preparation With Misoprostol Before Hysteroscopy: a Randomized Trial of Different Routes of Administration
Brief Title: Same-day Cervical Preparation With Misoprostol Before Hysteroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0083-15-WOMC
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Preparation Prior to Hysteroscopy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Care Provider

ARMS (3):
- PO Misoprostol (Active Comparator): Patients assigned to PO Misoprostol (Cytotec) 400 mg once, 2-4 hours prior to hysteroscopy
  Interventions: Drug: Misoprostol (Cytotec)
- PV Misoprostol (Active Comparator): Patients assigned to PV Misoprostol (Cytotec) 400 mg once, 2-4 hours prior to hysteroscopy
  Interventions: Drug: Misoprostol (Cytotec)
- Buccal Misoprostol (Active Comparator): Patients assigned to buccal Misoprostol (Cytotec) 400 mg once, 2-4 hours prior to hysteroscopy
  Interventions: Drug: Misoprostol (Cytotec)

INTERVENTIONS:
Drug: Misoprostol (Cytotec)

SUMMARY:
This is a randomized trial, assessing Misoprostol efficacy in cervical preparation several hours prior to hysteroscopy, comparing the different routes of administration (PO/PV/buccal). Initial cervical dilatation will be assessed, as well as surgical ease of dilatation, time required to achieve dilatation and patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective hysteroscopy (diagnostic/surgical) at Wolfson Medical Center
* Written consent supplied

Exclusion Criteria:

* Contraindications to prostaglandin treatment (severe asthma, glaucoma, severe cardiac disease, renal failure)
* Prostaglandin allergy
* Pregnancy
* Genital infection
* Space-occupying lesion in the endocervical canal
* Prior cervical surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Preoperative cervical width in centimeters | intraoperative
  Initial cervical dilatation assessed by performing cervical dilatation , beginning with a number 10 Hegar dilator and subsequently inserting smaller Hegar dilators until the dilator can pass through the internal os without resistance. The largest one to pass will consist the initial cervical width.

SECONDARY OUTCOMES:
Time required to achieve cervical dilatation | intraoperative
  The time in minutes required for dilatation up to a number 10 Hegar
Ease of cervical dilatation | intraoperative
  The subjective ease of cervical dilatation recorded by the surgeon on a 5-point Likert scale (1-very difficult, 5- very easy)
Patient preference | baseline
  Patient acceptability of the administration of medication on a 5-point Likert scale (1-very uncomfortable, 5-very comfortable)
Adverse effects of medication | baseline
  Self reported misoprostol-associated adverse effects before the procedure (such as nausea, vomiting)
Surgical complications | intraoperative
  Complications arising during surgery (perforation, cervical laceration, excess bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel

REFERENCES:
- [Derived] Ganer Herman H, Kerner R, Gluck O, Feit H, Keidar R, Bar J, Sagiv R. Different Routes of Misoprostol for Same-Day Cervical Priming Prior to Operative Hysteroscopy: A Randomized Blinded Trial. J Minim Invasive Gynecol. 2017 Mar-Apr;24(3):455-460. doi: 10.1016/j.jmig.2016.12.024. Epub 2017 Jan 7. PMID 28069480